CLINICAL TRIAL: NCT01284725
Title: Weaning of Immunosuppression in Nephritis of Lupus
Acronym: WIN-Lupus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-022859-30; 2010-15 (Other: AP HM)
Record Dates: First submitted 2011-01-21; First posted 2011-01-27 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Nephritis of Lupus
MeSH Terms: interventions — Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immunosuppressive treatment discontinuation, (Experimental)
  Interventions: Other: immunosuppressive treatment discontinuation
- Continuation of immunosuppressive therapy (Active Comparator): with MMF or AZA, with a background therapy with hydroxychloroquine, and possibly low-dose corticosteroids
  Interventions: Drug: mycophenolate mofetil or azathioprine

INTERVENTIONS:
Drug: mycophenolate mofetil or azathioprine
  Arms: Continuation of immunosuppressive therapy
Other: immunosuppressive treatment discontinuation
  Arms: immunosuppressive treatment discontinuation,

SUMMARY:
The investigators wish to evaluate the discontinuation of maintenance immunosuppressive treatment after 2 years in patients with stable remission after a proliferative lupus nephritis. The patients will be continuing their treatment with hydroxychloroquine, possibly associated with low dose corticosteroids.

DETAILED DESCRIPTION:
open multicenter randomized non-inferiority study, comparing 2 types of therapeutic strategies after 2 years of maintenance treatment:

* Group I: Continuation of immunosuppressive therapy with MMF or AZA, with a background therapy with hydroxychloroquine, and possibly low-dose corticosteroids.
* Group II: immunosuppressive treatment discontinuation, continuation of hydroxychloroquine, and possibly low-dose corticosteroids (15 mg / day).

ELIGIBILITY:
Inclusion Criteria:

* At least 18-years-old patient, woman or man,
* Patient having a lupus according to the criteria of the ACR,
* Patient having presented a glomérulonéphrite lupique proliférative (class III or IV Has +/-C, +/-list(classify) V) - first push or relapse - proved by renal biopsy,
* Patient having received for this push a treatment of attack by steroids with strong doses and cyclophosphamide or mycophénolate mofétil,
* Patient in the course of treatment of interview(maintenance) by azathioprine or mycophénolate mofétil for at least 2 years, and at most for 3 years, with at the time of the inclusion, mycophénolate mofétil? 1 gram / day or azathioprine? 50 in the daytime,
* Patient in reply renal complete or partial (criteria of the European, secondary consensus 2) since? 12 months,
* Patient under Plaquenil ® since? 6 months with a hydroxychloroquinémie = 750 µg / L,
* Patient having accepted of participated in the study and having signed a lit(enlightened) consent.

Exclusion Criteria:

* Patient presenting a severe chronic renal insufficiency (DFG estimated(esteemed) by MDRD < 30 ml / min / 1.73m ²),
* Patient having presented an extra-renal push having required an increase of corticoids à> 20 in the daytime during at least 7 days less than 6 months ago,
* Patient presenting a contraindication to the hydroxychloroquine,
* Unaffiliated patient in a national social security,
* Minor patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
discontinuation of maintenance immunosuppressive therapy | 2 years
  to demonstrate that discontinuation of maintenance immunosuppressive therapy does not expose patients to a greater risk of relapse of proliferative lupus nephritis compared to the continuation of this treatment

SECONDARY OUTCOMES:
compare 2 therapeutic strategies | 2 years
  to compare 2 therapeutic strategies in terms of relapse-free survival, overall survival , cumulative rate of 'relapse and / or death ', rates of adverse events , evolution of renal function , activity of SLE , consumption of steroids, impact on quality of life and economic impact.

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille; NOEMIE JOURDE CHICHE, Principal Investigator — Assistance publique Hôpitaux de marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Background] Himbert M, Jourde-Chiche N, Chapart L, Charles N, Baumstarck K, Daugas E. Anti-dsDNA IgE: a potential non-invasive test for prediction of lupus nephritis relapse. RMD Open. 2024 Jun 28;10(2):e004255. doi: 10.1136/rmdopen-2024-004255. PMID 38942591
- [Background] Jourde-Chiche N, Bobot M, Burtey S, Chiche L, Daugas E. Weaning Maintenance Therapy in Lupus Nephritis: For Whom, When, and How? Kidney Int Rep. 2023 May 22;8(8):1481-1488. doi: 10.1016/j.ekir.2023.05.012. eCollection 2023 Aug. PMID 37547513
- [Background] Jourde-Chiche N, Chiche L. An era of immunosuppressant withdrawal in systemic lupus erythematosus: winning through weaning. Lancet Rheumatol. 2024 Mar;6(3):e133-e134. doi: 10.1016/S2665-9913(24)00001-8. Epub 2024 Jan 29. No abstract available. PMID 38301681
- [Background] Chiche L, Jousse-Joulin S, Jourde-Chiche N. [From "Treat to Target" to "Think to Untreat": Therapeutic de-implementation as a new paradigm in systemic lupus erythematosus]. Rev Med Interne. 2023 Mar;44(3):101-104. doi: 10.1016/j.revmed.2022.12.001. Epub 2022 Dec 22. No abstract available. French. PMID 36566116
- [Result] Jourde-Chiche N, Costedoat-Chalumeau N, Baumstarck K, Loundou A, Bouillet L, Burtey S, Caudwell V, Chiche L, Couzi L, Daniel L, Deligny C, Dussol B, Faguer S, Gobert P, Gondran G, Huart A, Hummel A, Kalbacher E, Karras A, Lambert M, Le Guern V, Lebourg L, Loubiere S, Maillard-Lefebvre H, Maurier F, Pha M, Queyrel V, Remy P, Sarrot-Reynauld F, Verhelst D, Hachulla E, Amoura Z, Daugas E; WIN-Lupus study group. Weaning of maintenance immunosuppressive therapy in lupus nephritis (WIN-Lupus): results of a multicentre randomised controlled trial. Ann Rheum Dis. 2022 Oct;81(10):1420-1427. doi: 10.1136/annrheumdis-2022-222435. Epub 2022 Jun 20. PMID 35725295